CLINICAL TRIAL: NCT03799276
Title: Optimisation of Care and Antiretroviral Therapy in Vulnerable HIV Infected Individuals
Brief Title: Optimisation of Care in Vulnerable HIV Infected Individuals
Acronym: OPTICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Collaborators: ViiV Healthcare (Industry); Institut de Sante Publique, d'Epidemiologie et de Developpement (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CREPATS 08
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opticare study (Experimental): Phase I: Identification and Selection of study population The first step will include an active search by OPTICARE team for vulnerable and lost to follow up patients
  Phase II: Implementation of the individualized follow-up program The patients who agree to participate to the program will be defined as the OPTICARE population.
  Interventions: Other: Opticare study

INTERVENTIONS:
Other: Opticare study — Each patient will be evaluated by
  * An HIV physician
  * A nurse
  * A social worker
  * A psychological therapist
  * A cultural mediator/member of patients community if needed for migrants
  Following these interviews and visits, a multisciplinary team will define for each patient an individualized OPTICARE program based on the following items: clinical, psychological/psychiatric, social status and follow up visits will be planned with the patient.
  Regular (Day 15 and monthly) phone calls will be set up during the first six months of the OPTICARE program, to assess the clinical status and ART adherence.
  Patients will have their medical, biological and social status assessed through visits at W4, W12, W24, W36 (medical and social status only) and W 48 with all members of the OPTICARE team.

SUMMARY:
Antiretroviral therapy is currently the only way to control HIV disease progression in HIV infected subjects and to prevent transmission. However a sustained virological control through antiretroviral therapy is requested for these objectives. There is currently 8-10% of patients who failed therapy for many reasons other than virological resistance including social unstability, psychiatric disorders, migrant status, drug or alcohol addictions. Because many of these vulnerabilities can be managed and patients helped for following adequately cares and treatments, study team designed the OPTICARE Program to help reduce impact of the patients' vulnerabilities.

The OPTICARE study is designed as a prospective implementation interventional study which aims to improve retention in care among vulnerable HIV infected patients over 48 weeks.

The OPTICARE program is a support program dedicated to patients either lost to follow up or in highly fraility situation that will offer an individualized care management to fill their gaps towards optimized care and control of viral replication. Our aim is, in patients virally failing in relation with poor adherence to care and treatment to test first part whether tracking proactively lost to follow up patients or detecting frail individuals at risk of lost to care is effective and secondly to evaluate the efficacy, the feasibility and the acceptability of an intervention tailored to each individual to get them to treatment success with viral suppression. In our context, a randomized approach would not be seen as ethical or possible in an environment where investigators need to evaluate such intervention as a pilot approach. Investigators therefore enrolled patients in a cohort population study OPTICARE program aim to actively identify vulnerable HIV+ population and promote optimal access to health care to this population using retention in care program in order to enable long term HIV infection control.

The primary objective is to assess the feasability and the effectiveness of the OPTICARE program. The OPTICARE program aims to propose an individualized care to vulnerable HIV infected patients (UNAIDS/Second 90% goal) and to drive them to treatment success (UNAIDS/Third 90% goal) within a one-year period.

DETAILED DESCRIPTION:
The OPTICARE program is an individualized program proposed to vulnerable HIV infected patients according to a baseline evaluation of the clinical, social, psychological and cultural aspects.

Once enrolled in the OPTICARE program, each patient will benefit of:

* A comprehensive and complete check up personal interview, through a daily visit, with a physician, an educational nurse, a social worker and a cultural mediator (if needed), in order to identify mains issues
* A specific follow up will be set up with obligatory visits at week 4, week 12, week 24, week 36 and week 48 to assess the evolution of the previously identified issues. If needed, additional visits will be set up.
* Regular (Day 15 and monthly) phone calls will be set up during the first six months of the OPTICARE program.
* Each patient will be accompanied by a tutoring nurse who will be in direct contact with the patient.

Regarding the specific needs, each patient may benefit of:

* a personal assistance to complete administrative procedures (update health insurance, assistance to fill administrative papers, provide a budget for photo ID, transport tickets)
* a personalized medical follow up with regular phone calls, home visits (if the patient agrees), assistance in taking HIV medication (set up pillbox, therapeutic education)
* a close psychological and social support (connection with HIV organizations, participation to monthly support group)
* a specific assistance related to dependence issues (connection with addiction organization, sex therapist consultation)

A multidisciplinary team (physician, educational nurse, psychotherapist, social worker and cultural mediator) will proactively assist the patient (home visits, recall) during a one year follow up.

The program is initially proposed to the patient. In case of non-acceptance, the patient can further join the program after 3 months.

Patients who do not accept the OPTICARE program will be followed up in standard of care according to French HIV management guidelines. (https://cns.sante.fr/actualites/prise-en-charge-du-vih-recommandations-du-groupe-dexperts/). All administratives and social procedures will be given to the social district.

ELIGIBILITY:
Inclusion Criteria:

1. Patients Lost to follow-up defined as a patient with no clinical visit:

   * In the 12 months period for patients > 250/mm3 CD4 cells or
   * In the 6 months period for patients < 250/mm3 CD4 cells or
   * In the 3 months period following a new HIV + diagnosis or an AIDS defining illnesses

   AND with HIV plasma viral load > 400 cp/ml (following French HIV guidelines)
2. HIV+ patients with virological failure defined as HIV plasma viral load (pVL) > 400 cp/ml (2 determinations with at least two weeks apart)
3. HIV+ patients presenting with an AIDS defining (<3 months) event in a context of lost to care prior to the event
4. HIV+ patients newly diagnosed with virological failure 6 months after ART initiation (virological failure defined by two HIV plasma viral load > 50cp/ml following French HIV guidelines *) and with one of the following vulnerable risk factors :

   * Social frailty (lack of health insurance, homeless, accommodation by family/friends, post incarceration)
   * Migrants with a first arrival in France in the last 6 months
   * Women in postpartum period (3 months after delivery)
   * Psychiatric disease
   * Intravenous drug users, alcohol consumers (women > 40g/day or > 2 standard drinks /day; men > 60g/day ou > 3 standard drinks/day)

A standard glass is defined by a quantity of pure alcohol of 10 grams, corresponding to approximately 10 cl of wine, 25 cl of beer at 5% vol, or 3 cl of alcohol at 40% vol. (https://www.sfalcoologie.asso.fr/download/RBP2014-SFA-Mesusage-AA.pdf)

Exclusion Criteria:

* Patients unwilling to participate.
* Patients with HIV plasma viral load < 50 cp/ml

https://cns.sante.fr/actualites/prise-en-charge-du-vih-recommandations-du-groupe-dexperts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Measure of plasma viral load to assess the effectiveness of the OPTICARE Program to attend HIV plasma viral load < 50 cp/ml at week 48 | 12 months
  Measure of plasma viral load assessed by RNA quantification using COBAS 6800 system (Roche)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Seang, MD, Principal Investigator — Pitie Salpetriere Hospital
Locations (1):
- Yasmine Dudoit, Paris, France

IPD SHARING:
Plan to Share IPD: No